CLINICAL TRIAL: NCT03795935
Title: Relief From Side Effects: Clinical Use of Electrodes With Direction: a Prospective, Open Label, Clinical Trial for Thalamic Deep Brain Stimulation
Brief Title: Relief From Side Effects: Clinical Use of Electrodes With Direction
Acronym: RESCUED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Christopher Honey, Neurosurgeon, Professor of Surgery (Neurosurgery), Director of Surgical Centre for Movement Disorders, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H17-00672
Record Dates: First submitted 2018-09-17; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Deep Brain Stimulation; Directional Lead; Essential Tremor
Keywords: Deep Brain Stimulation; Directional Lead; Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients who were previously implanted with a traditional DBS lead and have subsequently developed stimulation induced side effects will gain significantly more tremor control without side effects when re-implanted with a directional DBS lead. We expect these patients' quality of life will improve. These patients typically will have had significant tremor relief (greater than 75% reduction from preoperative tremor rating scale) without side effects at their one year post operative follow-up. With the expected disease progression they will have had to increase their DBS stimulation to the degree that their DBS now causes side effects in order to block their tremor
  Interventions: Other: No side-effect stimulator settings with directional lead

INTERVENTIONS:
Other: No side-effect stimulator settings with directional lead — Individuals in this arm will have their stimulator settings programmed to the point in which they have maximum tremor control with no side effects.

SUMMARY:
Deep Brain Stimulation (DBS) uses electrical pulses sent through a lead (insulated wire) to help stop unwanted symptoms in a variety of brain diseases, including the tremor seen in patients with Essential Tremor (ET). The current standard lead allows this stimulation to spread out uniformly in all directions. As these diseases progress, however, the amount of electrical stimulation required to stop the symptom usually increases. This may become problematic because the increased electrical stimulation required for advanced symptoms may spread outside the desired targeted area, and effect other parts of the brain and causing unwanted side effects. A new type of DBS lead has been developed which can steer, or focus, the electrical stimulation in a given direction toward the desired target area and away from areas that would cause side effects. We would like to quantify the benefit seen in patients who have been switched from the traditional lead to this new directional lead.

DETAILED DESCRIPTION:
Patients implanted with a DBS may experience unwanted side effects such as motor contractures, paresthesia, or dysarthria. This occurs when the electrical field of the stimulation spreads out beyond the targeted area. This is especially common in patients whose disease has progressed, and must use increasingly higher currents in order to regain control of their tremor. Unfortunately, because the electrical field affects neurons in a symmetrical sphere around the DBS, it is often impossible to reach the additional desired neuronal elements without simultaneously affecting equidistant brain regions responsible for side effects. For many of our advanced patients, this means choosing between a debilitating tremor or disabling side effects.The directional lead is a FDA and Health Canada approved DBS lead which features radially segmented electrodes which can selectively steer the electrical field in a predefined direction, orthogonal to the lead trajectory. This will allow DBS clinicians to steer current towards desired structural areas, while avoiding locations, which produce negative side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been implanted with the DBS
* Participants must have been diagnosed with Essential Tremor
* Participants must experience negative side effects from their DBS which limit control over their tremor
* Participants must be able to receive benefit from their stimulator, but at the cost of negative side effects

Exclusion Criteria:

* All individuals who meet criteria outlined in "inclusion criteria" may be eligible for this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Tremor Control | Assessed once all tests performed - 1 to 2 months post-operatively
  Maximum percentage change in tremor (as measured by the Tremor Rating Scale) without side-effects (comparing DBS "on" versus "off") in each patient using the standard lead compared to the directional lead.

SECONDARY OUTCOMES:
Quality of life based on participant's best real life setting | Assessed during study visits - The initial assessment will occur during a pre-operative study visit which will be compared post operatively 3 months after outcome 1 has been measured
  Quality of life will be based on each participant's subjective opinion using the Short Form 36 (SF36) (a patient-reported survey focusing on health and quality of life) assessment form.
Quality of life based on tremor management participant's best real life setting | Assessed during study visits - The initial assessment will occur during a pre-operative study visit which will be compared post operatively 3 months after outcome 1 has been measured
  Quality of life will be based on each participant's subjective opinion using the Quality of Life in Essential Tremor Questionare.
Quality of life based on voice handicap with participant's best real life setting | Assessed during study visits - The initial assessment will occur during a pre-operative study visit which will be compared post operatively 3 months after outcome 1 has been measured
  Quality of life will be based on each participant's subjective opinion using the Vocal handicap Index scale.

CONTACTS AND LOCATIONS:
Locations (1):
- The Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toader E, Decre MM, Martens HC. Steering deep brain stimulation fields using a high resolution electrode array. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:2061-4. doi: 10.1109/IEMBS.2010.5626472. PMID 21096152
- [Background] Reinacher PC, Kruger MT, Coenen VA, Shah M, Roelz R, Jenkner C, Egger K. Determining the Orientation of Directional Deep Brain Stimulation Electrodes Using 3D Rotational Fluoroscopy. AJNR Am J Neuroradiol. 2017 Jun;38(6):1111-1116. doi: 10.3174/ajnr.A5153. Epub 2017 Apr 6. PMID 28385887